CLINICAL TRIAL: NCT04323397
Title: Nasal High Frequency Oscillatory Versus Synchronized Intermittent Positive Pressure Ventilation in Neonate Following Extubation: Randomized Controlled Crossover Study
Brief Title: Nasal HFOV Versus Nasal SIPPV in Neonate Following Extubation: RCT Crossover Study
Acronym: nHFOnSIPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Anucha Thatrimontrichai, Principal Investigator, Prince of Songkla University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 6238211
Record Dates: First submitted 2020-03-25; First posted 2020-03-26 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: High-Frequency Ventilation; Intermittent Positive-Pressure Ventilation; Newborn Morbidity; Noninvasive Ventilation
Keywords: Nasal High-Frequency Oscillation; Nasal Synchronized Intermittent Positive Pressure; Respiratory Failure; Extubation Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Crossover Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal high frequency oscillatory ventilation (Experimental): nHFO: flow 8-10 L/minute, frequency 10 Hz, MAP = "MAP (before extubation) + 2" or "8 (preterm), 10 (term)" cmH2O, dP = "2-3 times of MAP with visible chest oscillations" or 25-35 cmH2O, I:E = 1:1, FiO2 = "FiO2 (before extubation) + 0.1-0.2" keep targeted SpO2 90-94%
  Interventions: Device: Non-invasive ventilation
- nasal synchronized intermittent positive pressure ventilation (Experimental): nSIPPV: flow 8-10 L/minute, rate 60/minute, PIP = "PIP (before extubation) + 2-5" or "20 (preterm), 25 (term)" cmH2O, PEEP = 5 cmH2O, IT = 0.5 s, FiO2 = "FiO2 (before extubation) + 0.1-0.2" keep targeted SpO2 90-94%. The highest trigger sensitivity avoiding auto triggering was selected.
  Interventions: Device: Non-invasive ventilation

INTERVENTIONS:
Device: Non-invasive ventilation — Intervention nasal high frequency oscillatory ventilation (nHFOV) and nasal synchronized intermittent positive pressure ventilation (nSIPPV) were generated by neonatal ventilators (SLE6000 infant ventilators, United Kingdom) using bi-nasal prongs (RAM cannula, NEOTECH®, USA) or the nasal mask of the same type for both ventilation modes. The size of the prongs was determined by the infant's weight. The largest possible prongs were used, with a snug fit to avoid leakage. Pacifier for preterm and term neonate (Jollypop™, USA) was taken to avoid leakage from the mouth. The disposable ventilator circuit (Fisher & Paykel RT268™, Evaqua Dual Limb Infant Breathing Circuit Kit with Evaqua 2 Technology and Pressure Line, Flow > 4L/min, New Zealand) was used. The initial NIV setting was (7) described in arm description. (above)

SUMMARY:
Mechanical ventilation was introduced to treat respiratory failure in preterm infants or sick neonates then improvements in survival (1,2). However, the complications from short or long term use of ventilation can result in unintended harm or burden (e.g., air leak syndrome, pneumonia, bronchopulmonary dysplasia, neurological injury, retinopathy of prematurity) (3,4). To reduce these risks, clinicians should aggressive extubated neonates as early as possible. Respiratory (focus on blood gas as well as partial pressure CO2 [pCO2]) or extubation (focus on clinical condition as well as reintubation) failure was worrisome in pediatrician and parents if the neonate was reintubated owing to complete recovery of lung disease or inadequate respiratory drive.

Non-invasive ventilation (NIV) was supported for primary respiratory support (initial mode before endotracheal intubation) or post-extubation. Nasal continuous positive airway pressure (nCPAP) was familiar to NIV mode in neonatal respiratory support. Nowadays, the new NIV modalities are nasal intermittent synchronized positive pressure ventilation (nSIPPV) and nasal high frequency oscillation (nHFO). To increase the likelihood of nCPAP success, other new modalities of NIV may be interesting. From theory, nSIPPV and nHFO combines peak inspiratory pressure (PIP) with synchrony and high-frequency oscillations without synchrony above CPAP, respectively. From meta-analysis, nSIPPV and nHFO were statistically significant superior than nCPAP both respiratory and extubation failure in neonate (5,6).

The aim of our study was to investigate the efficacy of nHFOV and nSIPPV for CO2 clearance and reintubation rate after extubated neonates. The investigators hypothesized that nHFOV mode would improve CO2 clearance better than nSIPPV mode.

DETAILED DESCRIPTION:
The primary outcome (pCO2) was measured by crossover RCT. The secondary outcome (reintubation within 7 days) was measured by paralleled RCT.

ELIGIBILITY:
Inclusion Criteria:

* Born in hospital and admit in NICU
* The first endotracheal intubation and need NIV if extubation
* Umbilical arterial catheterization to draw the blood gas
* Neonate has not been intervened from another RCT study

Exclusion Criteria:

* Major congenital anomalies or chromosomal abnormalities
* Neuromuscular diseases
* Upper respiratory tract abnormalities
* Suspected congenital lung diseases or pulmonary hypoplasia
* Need for surgery known before the first extubation
* Grade IV intraventricular hemorrhage occurring before the first extubation
* Palliative care
* Parents' decision not to participate

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anucha Thatrimontrichai, M.D., Principal Investigator — Prince of Songkla University
Locations (1):
- Songklanagarind Hospital, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baingam K, Phatigomet M, Thatrimontrichai A, Maneenil G, Dissaneevate S, Janjindamai W. Carbon Dioxide Level between Nasal High-Frequency Oscillatory Ventilation and Synchronized Nasal Intermittent Positive Pressure Ventilation after Extubation in Neonates: A Cross-over Randomized Controlled Trial. Am J Perinatol. 2024 Aug;41(11):1495-1503. doi: 10.1055/a-2113-3284. Epub 2023 Jun 20. PMID 37339671
- [Result] Phatigomet M, Thatrimontrichai A, Maneenil G, Dissaneevate S, Janjindamai W. Reintubation Rate between Nasal High-Frequency Oscillatory Ventilation versus Synchronized Nasal Intermittent Positive Pressure Ventilation in Neonates: A Parallel Randomized Controlled Trial. Am J Perinatol. 2024 Aug;41(11):1504-1511. doi: 10.1055/a-2118-5351. Epub 2023 Jun 27. PMID 37369239
- [Result] Baingam K, Phatigomet M, Thatrimontrichai A, Maneenil G, Dissaneevate S, Janjindamai W. Erratum: Carbon Dioxide Level between Nasal High-Frequency Oscillatory Ventilation and Synchronized Nasal Intermittent Positive Pressure Ventilation after Extubation in Neonates: A Cross-over Randomized Controlled Trial. Am J Perinatol. 2024 Aug;41(11):e1. doi: 10.1055/s-0044-1778715. Epub 2024 Jan 24. No abstract available. PMID 38266755
- [Result] Phatigomet M, Thatrimontrichai A, Maneenil G, Dissaneevate S, Janjindamai W. Erratum: Reintubation Rate between Nasal High-Frequency Oscillatory Ventilation versus Synchronized Nasal Intermittent Positive Pressure Ventilation in Neonates: A Parallel Randomized Controlled Trial. Am J Perinatol. 2024 Aug;41(11):e2. doi: 10.1055/s-0044-1778714. Epub 2024 Jan 24. No abstract available. PMID 38266756

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 203 neonates were assessed for eligibility
Pre-assignment Details: The 133 participants were included in the study.
Groups:
- "nHFO First, Then nSIPPV, Then nHFO": nHFO: flow 8-10 L/minute, frequency 10 Hz, MAP = "MAP (before extubation) + 2" or "8 (preterm), 10 (term)" cmH2O, dP = "2-3 times of MAP with visible chest oscillations" or 25-35 cmH2O, I:E = 1:1, FiO2 = "FiO2 (before extubation) + 0.1-0.2" keep targeted SpO2 90-94%
  Non-invasive ventilation: Intervention nasal high frequency oscillatory ventilation (nHFOV) and nasal synchronized intermittent positive pressure ventilation (nSIPPV) were generated by neonatal ventilators (SLE6000 infant ventilators, United Kingdom) using bi-nasal prongs (RAM cannula, NEOTECH®, USA) or the nasal mask of the same type for both ventilation modes. The size of the prongs was determined by the infant's weight. The largest possible prongs were used, with a snug fit to avoid leakage. Pacifier for preterm and term neonate (Jollypop™, USA) was taken to avoid leakage from the mouth. The disposable ventilator circuit (Fisher & Paykel RT268™, Evaqua Dual Limb Infant Breathing Circuit Kit with Evaqua 2 Technology and Pressure Line, Flow > 4L/min, New Zealand) was used. The initial NIV setting was (7) described in arm description. (above)
- "nSIPPV First, Then nHFOV, Then nSIPPV": nSIPPV: flow 8-10 L/minute, rate 60/minute, PIP = "PIP (before extubation) + 2-5" or "20 (preterm), 25 (term)" cmH2O, PEEP = 5 cmH2O, IT = 0.5 s, FiO2 = "FiO2 (before extubation) + 0.1-0.2" keep targeted SpO2 90-94%. The highest trigger sensitivity avoiding auto triggering was selected.
  Non-invasive ventilation: Intervention nasal high frequency oscillatory ventilation (nHFOV) and nasal synchronized intermittent positive pressure ventilation (nSIPPV) were generated by neonatal ventilators (SLE6000 infant ventilators, United Kingdom) using bi-nasal prongs (RAM cannula, NEOTECH®, USA) or the nasal mask of the same type for both ventilation modes. The size of the prongs was determined by the infant's weight. The largest possible prongs were used, with a snug fit to avoid leakage. Pacifier for preterm and term neonate (Jollypop™, USA) was taken to avoid leakage from the mouth. The disposable ventilator circuit (Fisher & Paykel RT268™, Evaqua Dual Limb Infant Breathing Circuit Kit with Evaqua 2 Technology and Pressure Line, Flow > 4L/min, New Zealand) was used. The initial NIV setting was (7) described in arm description. (above)
Period: First Intervention
Arm/Group | "nHFO First, Then nSIPPV, Then nHFO" | "nSIPPV First, Then nHFOV, Then nSIPPV"
Started | 51 | 51
Completed | 51 (only neonates with arterial line) | 51 (only neonates with arterial line)
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | "nHFO First, Then nSIPPV, Then nHFO" | "nSIPPV First, Then nHFOV, Then nSIPPV"
Started | 51 | 51
Completed | 51 | 51
Not Completed | 0 | 0
Period: Third Intervention
Arm/Group | "nHFO First, Then nSIPPV, Then nHFO" | "nSIPPV First, Then nHFOV, Then nSIPPV"
Started | 67 (The participants, who were unavailable arterial line, were more enrolled and randomized to nHFO for 16 neonates (only the third intervention). Finally, the total participants were 67 (available arterial line and unavailable arterial line = 51 and 16, respectively)) | 66 (The participants, who were unavailable arterial line, were more enrolled and randomized to nSIPPV for 15 neonates (only the third intervention). Finally, the total participants were 66 (available arterial line and unavailable arterial line = 51 and 15, respectively))
Completed | 67 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- nHFOV, Then nSIPPV, Then nHFOV: nHFO: flow 8-10 L/minute, frequency 10 Hz, MAP = "MAP (before extubation) + 2" or "8 (preterm), 10 (term)" cmH2O, dP = "2-3 times of MAP with visible chest oscillations" or 25-35 cmH2O, I:E = 1:1, FiO2 = "FiO2 (before extubation) + 0.1-0.2" keep targeted SpO2 90-94%
  Non-invasive ventilation: Intervention nasal high frequency oscillatory ventilation (nHFOV) and nasal synchronized intermittent positive pressure ventilation (nSIPPV) were generated by neonatal ventilators (SLE6000 infant ventilators, United Kingdom) using bi-nasal prongs (RAM cannula, NEOTECH®, USA) or the nasal mask of the same type for both ventilation modes. The size of the prongs was determined by the infant's weight. The largest possible prongs were used, with a snug fit to avoid leakage. Pacifier for preterm and term neonate (Jollypop™, USA) was taken to avoid leakage from the mouth. The disposable ventilator circuit (Fisher & Paykel RT268™, Evaqua Dual Limb Infant Breathing Circuit Kit with Evaqua 2 Technology and Pressure Line, Flow > 4L/min, New Zealand) was used. The initial NIV setting was (7) described in arm description. (above)
- nSIPPV, Then nHFOV, Then nSIPPV: nSIPPV: flow 8-10 L/minute, rate 60/minute, PIP = "PIP (before extubation) + 2-5" or "20 (preterm), 25 (term)" cmH2O, PEEP = 5 cmH2O, IT = 0.5 s, FiO2 = "FiO2 (before extubation) + 0.1-0.2" keep targeted SpO2 90-94%. The highest trigger sensitivity avoiding auto triggering was selected.
  Non-invasive ventilation: Intervention nasal high frequency oscillatory ventilation (nHFOV) and nasal synchronized intermittent positive pressure ventilation (nSIPPV) were generated by neonatal ventilators (SLE6000 infant ventilators, United Kingdom) using bi-nasal prongs (RAM cannula, NEOTECH®, USA) or the nasal mask of the same type for both ventilation modes. The size of the prongs was determined by the infant's weight. The largest possible prongs were used, with a snug fit to avoid leakage. Pacifier for preterm and term neonate (Jollypop™, USA) was taken to avoid leakage from the mouth. The disposable ventilator circuit (Fisher & Paykel RT268™, Evaqua Dual Limb Infant Breathing Circuit Kit with Evaqua 2 Technology and Pressure Line, Flow > 4L/min, New Zealand) was used. The initial NIV setting was (7) described in arm description. (above)
- Total: Total of all reporting groups
Arm/Group | nHFOV, Then nSIPPV, Then nHFOV | nSIPPV, Then nHFOV, Then nSIPPV | Total
Number analyzed (Participants) | 67 | 66 | 133
Age, Continuous [Median (Inter-Quartile Range); unit: weeks] — Gestational age
  weeks | 33 [30 to 35] | 33 [30 to 37] | 33 [30 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 32 | 52
  Male | 47 | 34 | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Duration of invasive ventilation [Median (Inter-Quartile Range); unit: hours] | 63.4 [21.2 to 95.2] | 42.9 [21.7 to 84.1] | 48.4 [21.3 to 90.8]

OUTCOME MEASURES:

1. Primary Outcome: Partial Pressure CO2 (pCO2) : Data From the Crossover Phase of the Study
Description: Data from the Crossover Phase of the study: After randomization only in neonate with arterial line, the initial non-invasive ventilation (NIV) was started then blood gas was obtained after 2 hours. The participant was switched to another NIV and blood gas was obtained after 2 hours.
Time Frame: 2 hours after each intervention
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- nHFO: nHFO: flow 8-10 L/minute, frequency 10 Hz, MAP = "MAP (before extubation) + 2" or "8 (preterm), 10 (term)" cmH2O, dP = "2-3 times of MAP with visible chest oscillations" or 25-35 cmH2O, I:E = 1:1, FiO2 = "FiO2 (before extubation) + 0.1-0.2" keep targeted SpO2 90-94%
  Non-invasive ventilation: Intervention nasal high frequency oscillatory ventilation (nHFOV) and nasal synchronized intermittent positive pressure ventilation (nSIPPV) were generated by neonatal ventilators (SLE6000 infant ventilators, United Kingdom) using bi-nasal prongs (RAM cannula, NEOTECH®, USA) or the nasal mask of the same type for both ventilation modes. The size of the prongs was determined by the infant's weight. The largest possible prongs were used, with a snug fit to avoid leakage. Pacifier for preterm and term neonate (Jollypop™, USA) was taken to avoid leakage from the mouth. The disposable ventilator circuit (Fisher & Paykel RT268™, Evaqua Dual Limb Infant Breathing Circuit Kit with Evaqua 2 Technology and Pressure Line, Flow > 4L/min, New Zealand) was used. The initial NIV setting was (7) described in arm description. (above)
- nSIPPV: nSIPPV: flow 8-10 L/minute, rate 60/minute, PIP = "PIP (before extubation) + 2-5" or "20 (preterm), 25 (term)" cmH2O, PEEP = 5 cmH2O, IT = 0.5 s, FiO2 = "FiO2 (before extubation) + 0.1-0.2" keep targeted SpO2 90-94%. The highest trigger sensitivity avoiding auto triggering was selected.
  Non-invasive ventilation: Intervention nasal high frequency oscillatory ventilation (nHFOV) and nasal synchronized intermittent positive pressure ventilation (nSIPPV) were generated by neonatal ventilators (SLE6000 infant ventilators, United Kingdom) using bi-nasal prongs (RAM cannula, NEOTECH®, USA) or the nasal mask of the same type for both ventilation modes. The size of the prongs was determined by the infant's weight. The largest possible prongs were used, with a snug fit to avoid leakage. Pacifier for preterm and term neonate (Jollypop™, USA) was taken to avoid leakage from the mouth. The disposable ventilator circuit (Fisher & Paykel RT268™, Evaqua Dual Limb Infant Breathing Circuit Kit with Evaqua 2 Technology and Pressure Line, Flow > 4L/min, New Zealand) was used. The initial NIV setting was (7) described in arm description. (above)
Arm/Group | nHFO | nSIPPV
Number analyzed (Participants) | 102 | 102
mm Hg | 38.7 (8.8) | 36.8 (10.2)

2. Secondary Outcome: Number of Participants With Extubation Failure: Data From the Parallel Phase of the Study.
Description: Data from the Parallel Phase of the study: The participant with and without arterial line was randomized. If The participant with arterial line was randomized to cross-over trial (randomized to NIV, then switched to another NIV for 2 hours, then switched to the first NIV [parallel trial]). If The participant without arterial line was randomized to parallel trial. Extubation failure will be defined by reintubation after NIV mode.
Time Frame: up to 7 days after each intervention
Measure: Count of Participants; unit: Participants
Arm/Group | nHFO | nSIPPV
Number analyzed (Participants) | 67 | 66
Participants | 5 | 4

ADVERSE EVENTS:
Time Frame: Adverse event: "Crossover Phase: up to 4 hours, Parallel Phase: up to 7 days after intervention"
Description: "Crossover Phase: up to 6 hours (participants = 51 neonate, 102 periods each arm for crossover), Parallel Phase: up to 7 days after intervention (participants = 67+66 = 133 participants)"
Groups:
- Parallel: Nasal High Frequency Oscillatory Ventilation: nHFO: flow 8-10 L/minute, frequency 10 Hz, MAP = "MAP (before extubation) + 2" or "8 (preterm), 10 (term)" cmH2O, dP = "2-3 times of MAP with visible chest oscillations" or 25-35 cmH2O, I:E = 1:1, FiO2 = "FiO2 (before extubation) + 0.1-0.2" keep targeted SpO2 90-94%
  Non-invasive ventilation: Intervention nasal high frequency oscillatory ventilation (nHFOV) and nasal synchronized intermittent positive pressure ventilation (nSIPPV) were generated by neonatal ventilators (SLE6000 infant ventilators, United Kingdom) using bi-nasal prongs (RAM cannula, NEOTECH®, USA) or the nasal mask of the same type for both ventilation modes. The size of the prongs was determined by the infant's weight. The largest possible prongs were used, with a snug fit to avoid leakage. Pacifier for preterm and term neonate (Jollypop™, USA) was taken to avoid leakage from the mouth. The disposable ventilator circuit (Fisher & Paykel RT268™, Evaqua Dual Limb Infant Breathing Circuit Kit with Evaqua 2 Technology and Pressure Line, Flow > 4L/min, New Zealand) was used. The initial NIV setting was (7) described in arm description. (above)
- Parallel: Nasal Synchronized Intermittent Positive Pressure Ventilation: nSIPPV: flow 8-10 L/minute, rate 60/minute, PIP = "PIP (before extubation) + 2-5" or "20 (preterm), 25 (term)" cmH2O, PEEP = 5 cmH2O, IT = 0.5 s, FiO2 = "FiO2 (before extubation) + 0.1-0.2" keep targeted SpO2 90-94%. The highest trigger sensitivity avoiding auto triggering was selected.
  Non-invasive ventilation: Intervention nasal high frequency oscillatory ventilation (nHFOV) and nasal synchronized intermittent positive pressure ventilation (nSIPPV) were generated by neonatal ventilators (SLE6000 infant ventilators, United Kingdom) using bi-nasal prongs (RAM cannula, NEOTECH®, USA) or the nasal mask of the same type for both ventilation modes. The size of the prongs was determined by the infant's weight. The largest possible prongs were used, with a snug fit to avoid leakage. Pacifier for preterm and term neonate (Jollypop™, USA) was taken to avoid leakage from the mouth. The disposable ventilator circuit (Fisher & Paykel RT268™, Evaqua Dual Limb Infant Breathing Circuit Kit with Evaqua 2 Technology and Pressure Line, Flow > 4L/min, New Zealand) was used. The initial NIV setting was (7) described in arm description. (above)
- Crossover: Nasal High Frequency Oscillatory Ventilation: nHFO: flow 8-10 L/minute, frequency 10 Hz, MAP = "MAP (before extubation) + 2" or "8 (preterm), 10 (term)" cmH2O, dP = "2-3 times of MAP with visible chest oscillations" or 25-35 cmH2O, I:E = 1:1, FiO2 = "FiO2 (before extubation) + 0.1-0.2" keep targeted SpO2 90-94%
- Crossover: Nasal Synchronized Intermittent Positive Pressure Ventilation: nSIPPV: flow 8-10 L/minute, rate 60/minute, PIP = "PIP (before extubation) + 2-5" or "20 (preterm), 25 (term)" cmH2O, PEEP = 5 cmH2O, IT = 0.5 s, FiO2 = "FiO2 (before extubation) + 0.1-0.2" keep targeted SpO2 90-94%. The highest trigger sensitivity avoiding auto triggering was selected.
Arm/Group | Parallel: Nasal High Frequency Oscillatory Ventilation | Parallel: Nasal Synchronized Intermittent Positive Pressure Ventilation | Crossover: Nasal High Frequency Oscillatory Ventilation | Crossover: Nasal Synchronized Intermittent Positive Pressure Ventilation
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/66 | 0/102 | 0/102
Serious Adverse Events (participants affected / at risk) | 5/67 | 4/66 | 0/102 | 1/102
Other Adverse Events (participants affected / at risk) | 0/67 | 0/66 | 0/102 | 0/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parallel: Nasal High Frequency Oscillatory Ventilation (N=67) | Parallel: Nasal Synchronized Intermittent Positive Pressure Ventilation (N=66) | Crossover: Nasal High Frequency Oscillatory Ventilation (N=102) | Crossover: Nasal Synchronized Intermittent Positive Pressure Ventilation (N=102)
Adverse Event after started intervention (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 0 (0) | 1 (1) — Reintubation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT04323397/Prot_SAP_000.pdf